CLINICAL TRIAL: NCT00754507
Title: Efficacy of WelChol as an Add-on to Atorvastatin Therapy
Brief Title: A Study to Determine the Effect of WelChol Tablets on Cholesterol in Patients Who Have Been Taking Atorvastatin for at Least 4 Weeks.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Senior Director of Metabolic Research, Daiichi Sankyo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-406
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): colesevelam tablets and atorvastatin tablets
  Interventions: Drug: colesevelam HCl tablets, and atorvastatin tablets
- 2 (Placebo Comparator): colesevelam HCl placebo tablets and atorvastatin tablets
  Interventions: Drug: colesevelam HCl placebo tablets and atorvastatin tablets

INTERVENTIONS:
Drug: colesevelam HCl tablets, and atorvastatin tablets — colesevelam HCl tablets,6 tablets/day; atorvastatin tablets, 1 tablets/day for 6 weeks
  Arms: 1
Drug: colesevelam HCl placebo tablets and atorvastatin tablets — colesevelam HCl placebo tablets, 6 tablets/day for 6 weeks atorvastatin tablets, 1 tablet/day for 6 weeks
  Arms: 2

SUMMARY:
To determine the effects of WelChol tablets on serum lipids, lipoproteins, apolipoproteins, and lipoprotein particle size in patients who were stabilized on atorvastatin therapy for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > or greater than 18 years of age
* On a stable dose of atorvastatin
* LDL-C > or = to 115 mg/dL and < or = to 250 mg/dL
* TG < or = to 300 mg/dL
* Women are not pregnant or breast-feeding or planning to become pregnant
* Women of child-bearing potential had a hysterectomy or tubal-ligation, or
* women were post menopausal, or
* women practiced an acceptable method of contraception as specified in the protocol

Exclusion Criteria:

* BMI > 40 kg/m2
* History of allergic or toxic reaction to colesevelam HCl
* History of swallowing disorders
* Any serious disorder that could impact the conduct of the study
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the percent change in LDL-C from baseline to endpoint. | 6 weeks

SECONDARY OUTCOMES:
The absolute change in LDL-C from baseline to endpoint | 6 weeks
The absolute change and % change in total cholesterol | 6 Weeks
The absolute change and % change in triglycerides | 6 Weeks
The absolute change and % change in HDL-C | 6 Weeks
The absolute change and % change in C-reactive protein | 6 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Los Angeles, California
  - Castle Rock, Colorado
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Indianapolis, Indiana
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Bartlett, Tennessee
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington